CLINICAL TRIAL: NCT05417516
Title: A Randomized Trial of Five-Fraction Partial Breast Irradiation (RAPID2)
Brief Title: A Randomized Trial of Five Fraction Partial Breast Irradiation (RAPID2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCOG-2022-RAPID2
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm Female; Radiotherapy; Cosmetic Outcome

STUDY DESIGN:
Who Masked: Participant
Masking Description: Study participants will be made unaware of treatment allocation to prevent any potential bias in their assessment of cosmesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Breast Irradiation (WBI) (Active Comparator): 26 Gy in 5 fractions to the whole breast
  Interventions: Radiation: Whole Breast Irradiation (WBI)
- Partial Breast Irradiation (PBI) (Experimental): 26 Gy in 5 fractions to the tumour bed with a margin of normal tissue
  Interventions: Radiation: Partial Breast Irradiation (PBI)

INTERVENTIONS:
Radiation: Whole Breast Irradiation (WBI) — The dose fractionation and prescription is 26Gy in 5 fractions to the PTV once per day over 5-7 days (due to holiday weekends up to 8 days will be acceptable).
  Arms: Whole Breast Irradiation (WBI)
Radiation: Partial Breast Irradiation (PBI) — The dose fractionation and prescription is 26Gy in 5 fractions to the PTV prescribed at the isocentre of the treatment fields treated once per day over 5-7 days (due to holiday weekends up to 8 days will be acceptable).
  Arms: Partial Breast Irradiation (PBI)

SUMMARY:
The primary objective of this study is to determine in women with node negative BC ≤3cm in size, if PBI compared to WBI, both given once-a-day over 1 week following BCS, is non-inferior for LR and reduces adverse cosmesis. The primary outcomes are LR and patient-assessed cosmesis at 3 years post randomization.

DETAILED DESCRIPTION:
This is a randomized, two-arm, single blinded trial comparing two radiation treatment modalities, PBI and WBI. Following BCS or on the completion of additional adjuvant chemotherapy, eligible and consenting patients with newly diagnosed and histologically confirmed invasive carcinoma of the breast (without evidence of metastatic disease); with microscopically clear resection margins of 1mm (or no residual disease on re-excision) and negative axillary node involvement will be randomized in a 1:1 fashion to receive either PBI (experimental group) or WBI (control group). Study participants will receive 26Gy in 5 fractions in both treatment arms, treated once per day, for a period of 5-7 days. Study participants will not be made aware of treatment allocation to prevent any potential bias in their assessment of cosmesis. Stratification factors include tumour size, estrogen receptor (ER) status, and clinical centre.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in this study, patients must fulfill all of the following criteria:

1. Female with a new histological diagnosis of invasive carcinoma of the breast with no evidence of metastatic disease (see AJCC TNM Cancer Staging, Appendix II).
2. Treated by BCS with microscopically clear resection margins >= 1mm for invasive and non-invasive disease or no residual disease on re-excision.
3. Negative axillary node involvement as determined by either sentinel lymph node biopsy or axillary node dissection or clinical assessment with a negative axillary ultrasound and/or biopsy, for women with unifocal tumours <= 2cm, histologic grade 1 or 2, ER or PR+ and HER2-ve that are being planned for endocrine therapy

Exclusion Criteria:

Patients who satisfy any of the following exclusion criteria are NOT eligible for this study:

1. Age less than 50 years.
2. Known to be BRCA 1 and/or BRCA 2 positive.
3. Tumour size >3cm in greatest diameter on pathological examination.
4. Evidence of extensive intraductal component (EIC) (defined as an invasive tumour with a ductal carcinoma in situ (DCIS) component comprising at least 25% and extending beyond the invasive component to surrounding normal breast tissue) with the following exception: smaller tumours with EIC where the combined size (of the invasive and DCIS components) are <= 3cm remain eligible
5. Evidence of a DCIS component > 3cm
6. Lobular carcinoma only.
7. More than one primary tumour in different quadrants of the same breast (patients with multifocal breast cancer are eligible).
8. Synchronous or previous contralateral breast cancer (patients with contralateral DCIS or LCIS are eligible).
9. History of non-breast malignancy within the last 5 years other than treated non-melanoma skin cancer or treated in-situ carcinoma.
10. Known pregnancy or currently lactating.
11. Inability to localize tumour bed on CT planning (no evidence of surgical clips or seroma).
12. Inability to plan the patient for the experimental technique.

Ages: 50 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Local Recurrence | Annually for 5 years post-randomization
  Time from randomization to any evidence of tumour recurrence (invasive and non-invasive) in the treated breast.
Patient Assessment Cosmesis at 3 years | 3 and 5 years post-randomization
  Cosmesis will be assessed by the patient using the Breast Cosmesis Questionnaire which incorporates the Modified EORTC Breast Cosmetic Rating System and the UK Patient Reported Outcomes Questions following BCS.

SECONDARY OUTCOMES:
Distant Disease Free Survival (DDSF) | Annually for 5 years post-randomization.
  Time from randomization to evidence of metastasis involving distant sites (e.g. bone, liver, lung, or brain).
Disease Free Survival (DFS) | Annually for 5 years post-randomization.
  Time from randomization to local recurrence, regional or distant recurrence, contralateral breast cancer, other second cancer, or death.
Overall Survival | 3 years post-randomizaton.
  Time from randomization to death of any cause.
Radiation Toxicity | 2 weeks and 3 months post-radiation treatment, then annually for 5 years post-randomization.
  Acute (2 weeks and up to 3 months after completing RT) and late toxicity (beyond the 3 months after completing RT) will be assessed by clinical centre personnel using the NCI CTCAE version 5.0.
Nurse/Clinical Research Associate assessed cosmesis at 3 and 5 years. | 3 and 5 years post-randomization.
  A nurse/Clinical Research Associate (CRA) assessment of cosmesis using the EORTC Breast Cosmetic Rating System. Nurses and CRAs will be training in assessing cosmesis using training slides and guide previously developed for other trials.
Patient Assessed Cosmesis at 5 years. | 5 years post-randomization.
  Cosmesis will be assessed by the patient using the Breast Cosmesis Questionnaire which incorporates the Modified EORTC Breast Cosmetic Rating System13,27,42 and the UK Patient Reported Outcomes Questions following BCS.
Patient Reported Quality of Life | 2 weeks post-radiation treatment, then at 3 and 5 years post-randomization.
  Patients will complete the EORTC Breast Cancer Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Whelan, M.D., Principal Investigator — Juravinski Cancer Centre and McMaster University
Locations (26):
- Australia (10):
  - GenesisCare Hurstville, Hurstville, New South Wales
  - GenesisCare Mater Hospital, North Sydney, New South Wales
  - GenesisCare Bundaberg, Bundaberg, Queensland
  - GenesisCare Southport, Southport, Queensland
  - GenesisCare Tugun, Tugun, Queensland
  - GenesisCare Hervey Bay, Urraween, Queensland
  - GenesisCare St Andrew's, Adelaide, South Australia
  - GenesisCare Wembley, Wembley, Washington
  - GenesisCare Fiona Stanley Hospital, Murdoch, Western Austrailia
  - GenesisCare Hollywood, Nedlands, Western Australia
- Canada (16):
  - Arthur J. E. Child Comprehensive Cancer Centre-Clinical Research Unit, Calgary, Alberta
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - QEII HSC - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Stronach (Southlake) Regional Health Centre, Newmarket, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Toronto-Sunnybrook Health Sciences Centre - Odette Cancer Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CSSS Champlain - Charles LeMoyne, Greenfield Park, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux de la Mauricie-Centre-du-Québec (CIUSSS MCQ), Trois-Rivières, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No